CLINICAL TRIAL: NCT02146963
Title: Study of the BDNF- Val66Met Polymorphism in Alcohol-dependent Subjects in Relation to Abstinence After Withdrawal
Brief Title: Study of the BDNF-Val66Met Polymorphism in Alcohol-dependent Subjects in Relation to Abstinence After Withdrawal
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Philippe Nubukpo, MD, PhD, Centre Hospitalier Esquirol
Other Study IDs: 2014-A00613-44
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- alcohol withdrawal

SUMMARY:
This study is complementary to the main study "Brain Derived Neurotrophic Factor Serum Levels Evolution During the Six Months After Alcohol Withdrawal " NCT01491347.

The purpose of this study is to evaluate the Bdnf gene - Val66Met polymorphism in subjects with alcohol dependence according to their alcohol consumption status 6 months after withdrawal (relapse or abstinence), in relation to the presence of psychiatric co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* participation to the study "BDNF serum levels evolution during 6 months after alcohol withdrawal" (main study)
* criteria from the main study

Exclusion Criteria:

* criteria from the main study
* released or out from the main study before the follow-up at 4 months after withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: alcohol-dependent subjects hospitalized for alcohol withdrawal
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Frequency of the Bdnf gene Val/Val, Val/Met and Met/Met phenotypes as a function of relapse | at the time of inclusion

SECONDARY OUTCOMES:
serum BDNF levels variations between inclusion and 6 months later (or 4 months if the participants does not come for the 4 months-follow-up). | 6 months after alcohol withdrawal
existence of a psychiatric co-morbidity at the inclusion (major depression, schizophrenia, anxiety disorder) | at the time of inclusion
presence of a psychiatric co-morbidity at 6 months after withdrawal (major depression, schizophrenia, anxiety disorder) | 6 month after alcohol withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nubukpo, MD, PhD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France